CLINICAL TRIAL: NCT04324021
Title: A Phase 2/3, Randomized, Open-label, Parallel Group, 3-arm, Multicenter Study Investigating the Efficacy and Safety of Intravenous Administrations of Emapalumab, an Anti-interferon Gamma (Anti-IFNγ) Monoclonal Antibody, and Anakinra, an Interleukin-1(IL-1) Receptor Antagonist, Versus Standard of Care, in Reducing Hyper-inflammation and Respiratory Distress in Patients With SARS-CoV-2 Infection.
Brief Title: Efficacy and Safety of Emapalumab and Anakinra in Reducing Hyperinflammation and Respiratory Distress in Patients With COVID-19 Infection.
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Standard of care evolved during the timeframe of the study and had critical impact on recruitment.
  Early termination was not based on safety reasons but due to the reasons mentoined above.
  The ongoing patients were completed.
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sobi.IMMUNO-101; 2020-001167-93 (EudraCT Number)
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Results first posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: SARS-CoV-2
MeSH Terms: interventions — Emapalumab; Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Emapalumab (Active Comparator): Emapalumab i.v. infusion every 3rd day for a total 5 infusions. Day 1: 6mg/kg. Days 4, 7, 10 and 13: 3 mg/kg
  Interventions: Biological: Emapalumab
- Anakinra (Active Comparator): Anakinra i.v. infusion four times daily for 15 days. 400 mg/day in total, divided into 4 doses given every 6 hours
  Interventions: Biological: Anakinra
- Standard of care (No Intervention): Standard of care according to local practice

INTERVENTIONS:
Biological: Emapalumab — I.v. infusion every third day
  Other Names: Gamifant
  Arms: Emapalumab
Biological: Anakinra — Daily i.v. infusion
  Other Names: Kineret
  Arms: Anakinra

SUMMARY:
Hyper-inflammation, caused by a cytokine storm resulting from an exaggerated response of the immune system in the presence of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), is considered to represent one of the most important negative prognostic factors in patients infected with sSARS-CoV-2. The objective of this study is to investigate new treatment options to reduce the number of patients requiring mechanical ventilation. This is intended to address the most urgent need to preserve the access to intensive care unit support to the lowest possible number of patients and may potentially reduce mortality.

DETAILED DESCRIPTION:
This is an open label, controlled, parallel group, 3-arm, multicenter study to assess the efficacy and safety of Emapalumab or Anakinra, versus standard of care (SoC). Patients between 30 and 80 years will be eligible to participate in the study. The study is planned to consist of three groups, each comprising 18 patients. Treatment will be randomized to either Emapalumab+SoC, Anakinra+SoC or only SoC for two weeks. Follow-up visit or phone calls will be made 4 and 8 weeks after end of treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent provided by the patient, or by the patient's legally authorized representative(s), as applicable.
2. Documented presence of SARS-CoV-2 infection as per hospital routine.
3. Age > 18 to < 85 years at the time of screening.
4. Presence of respiratory distress, defined as:

   1. PaO2/FiO2 < 300 mm Hg and >200 mm Hg or
   2. Respiratory Rate (RR) ≥30 breaths/min or
   3. SpO2 < 93 percent in air at rest. Note: Patients given continous positive airway pressure (CPAP) ventilator support are eligible for inclusion.

Presence of hyperinflammation defined as:

1. Lymphocyte counts:

   * < 1000 cells/µL, in patients who have not received systemic glucocorticoids for at least 2 days prior to the assessment of the lymphocyte count
   * < 1200 cells/µL, in patients who have received systemic glucocorticoids for at least 2 days prior to the assessment of the lymphocyte count

   and
2. One of the following three criteria:

i. Ferritin > 500ng/mL

ii. LDH > 300 U/L

iii. D-Dimers > 1000 ng/mL

Exclusion Criteria:

1. Patients in mechanical ventilation or with modified early warning score (MEWS) >4 with evidence of moderate or above ARDS (Berlin definition, namely with PaO2/FiO2 >100, but <200 mm Hg) or severe respiratory insufficiency or evidence of rapid worsening (respiratory distress requiring mechanical ventilation or presence of shock or presence of concomitant organ failure requiring ICU admission). Note: For the evaluation of patient eligibility, temperature will not be considered in the calculation of the total MEWS score since presence of fever is a hallmark of SARS-CoV-2 infection
2. Impairment of cardiac function defined as poorly controlled heart diseases, such as New York heart association (NYHA) class II (mild) and above, cardiac insufficiency, unstable angina pectoris, myocardial infarction within 1 year before enrollment, supraventricular or ventricular arrhythmia need treatment or intervention.
3. Severe renal dysfunction (estimated glomerular filtration rate ≤ 30 mL/min/1.73 m2) or receive continuous renal replacement therapy, hemodialysis, or peritoneal dialysis.
4. Uncontrolled hypertension (seated systolic blood pressure >180 mmHg, or diastolic blood pressure >110mmHg) .
5. Administration of plasma from convalescent patients who recovered from SARS-CoV-2 infection.
6. Clinical suspicion of latent tuberculosis.
7. History of hypersensitivity or allergy to any component of the study drug.
8. Pregnant women.
9. Existence of any life-threatening co-morbidity or any other medical condition which, in the opinion of the investigator, makes the patient unsuitable for inclusion.
10. Enrollment in another concurrent clinical interventional study, or intake of an investigational drug within three months or 5 half-lives prior to inclusion in this study, if considered interfering with this study objectives as assessed by the Investigator.
11. Foreseeable inability to cooperate with given instructions or study procedures.
12. Clinical suspicion of active mycobacteria, histoplasma capsulatum, herpes zoster, salmonella, and shigella Infections.
13. Patients with liver dysfunction defined as AST or ALT > 5 × ULN

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Nicastri, MD, Principal Investigator — Direttore Dipartimento di Malattie Infettive
Locations (12):
- United States (5):
  - Regions hospital, Saint Paul, Minnesota
  - The Valley hospital, Ridgewood, New Jersey
  - NewYork-Presbyterian Queens, Flushing, New York
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Utah Health, Salt Lake City, Utah
- Italy (7):
  - ASST Spedali Civili di Brescia Dipartimento di Reumatologia e Immunologia Clinica, Brescia
  - S.C. Malattie Infettive, Ospedale Galliera, Genova
  - Ospedale Maggiore Policlinico, Dipartimento di Anestesia-Rianimazione e Medicina di Urgenza, Milan
  - Dipartimento di Medicina - DIMED, Azienda Ospedale - Università Padova, Padua
  - Azienda Ospedaliero-Universitaria di Parma, Dipartimento di Malattie infettive ed epatologia, Parma
  - Ospedale Lazzaro Spallanzani, Dipartimento di Malattie Infettive ad alta Intensità di cura ed altamente contagiose,Ospedale Lazzaro Spallanzani, Roma
  - ASL Città di Torino, Unit of Infectious Diseases, Medicine, Rheumatology, Torino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brands X, de Vries FMC, Uhel F, Haak BW, Peters-Sengers H, Schuurman AR, van Engelen TSR, Lutter R, Cremer OL, Bonten MJ, Schultz MJ, Scicluna BP, van der Poll T; MARS Consortium. Plasma Ferritin as Marker of Macrophage Activation-Like Syndrome in Critically Ill Patients With Community-Acquired Pneumonia. Crit Care Med. 2021 Nov 1;49(11):1901-1911. doi: 10.1097/CCM.0000000000005072. PMID 33935163

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were screened within 72h prior to the first IMP administration. A total of 54 patients were planned to be randomized. A total of 16 patients were randomized and analyzed.
Period: Overall Study
Arm/Group | Emapalumab | Anakinra | Standard of Care
Started | 5 | 5 | 6
Completed | 3 | 4 | 5
Not Completed | 2 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Death | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Emapalumab | Anakinra | Standard of Care | Total
Number analyzed (Participants) | 5 | 5 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (14.8) | 62.4 (11.1) | 62.5 (62.5) | 63.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2
  Male | 4 | 4 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 4 | 3 | 5 | 12
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Italy | 5 | 5 | 6 | 16
Hospitalization [Count of Participants; unit: Participants] | 5 | 5 | 6 | 16
Height (cm) [Mean (Standard Deviation); unit: cm] — Population: Data not available for the whole population
  cm
    number analyzed (Participants) | 5 | 5 | 4 | 14
    (all) | 170.8 (10.9) | 170.2 (4.4) | 172.3 (14.4) | 171 (9.5)
Weight (kg) [Mean (Standard Deviation); unit: kg] — Population: Data not available for the whole population
  kg
    number analyzed (Participants) | 5 | 5 | 4 | 14
    (all) | 77.4 (15.0) | 79.4 (13.4) | 83.0 (12.8) | 79.7 (13)
Symptom duration (days) [Mean (Standard Deviation); unit: days] — Screening date - disease symptom onset date + 1. If only year and month is present for symptom onset, the 15th of the month is used. If only year is present, June 30th is used.
  days | 4.0 (4.2) | 1.0 (0) | 5.3 (4.8) | 3.6 (4.0)
Oxygen levels (mmHg) [Mean (Standard Deviation); unit: mmHg] — Population: Data not available for the whole population
  mmHg
    number analyzed (Participants) | 4 | 4 | 5 | 13
    (all) | 103.0 (38.2) | 78.5 (21.0) | 78.6 (20.5) | 85.2 (27.7)
Fraction of Inspired oxygen (FiO2) (%) [Mean (Standard Deviation); unit: % of inspired oxygen] — Population: Data not available for the whole population
  % of inspired oxygen
    number analyzed (Participants) | 4 | 4 | 5 | 13
    (all) | 61.8 (29.9) | 54.8 (37.1) | 53.2 (22.4) | 56.3 (27.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Success
Description: Defined as the number of patients not requiring invasive mechanical ventilation or Extracorporeal membrane oxygenation (ECMO)
Time Frame: Up to Day 15
Measure: Count of Participants; unit: Participants
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
Participants | 3 | 4 | 5

2. Secondary Outcome: Number of Participants Requiring Mechanical Ventilation
Description: Measured in number of participants
Time Frame: Date of randomization to date of mechanical ventilation, up to 15 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
Participants | 1 | 1 | 1

3. Secondary Outcome: Change From Baseline in Modified Early Warning System Score
Description: The full (unabbreviated) scale name is Modified Early Warning system score (MEWS score) Measured in total score Total score is the sum of 5 categorized components (blood pressure, heart rate, respiratory rate, temperature and alert/voice/pain/unresponsive score) that are assigned a score between 0 and 2 or 0 and 3.
  MEWS total score range is 0 to 14. Higher score= worse outcome
Time Frame: Baseline, Day 15
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
scores on a scale | -1.00 (0.00) | 0.00 (0.82) | -0.75 (0.96)

4. Secondary Outcome: Change From Baseline in Ferritin
Description: Measured in local units
Time Frame: Baseline, Days 4, 7, 10, 13 and 15
Population: Change from baseline at Days 4, 7, 10, 13 and 15 Data not available for all patients at all timepoints
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
pmol/L
  Change from Baseline at D4: number analyzed (Participants) | 5 | 3 | 5
  Change from Baseline at D4 | -380.8 (3026.3) | -2864.2 (3789.3) | -770.2 (1093.0)
  Change from Baselind at D7: number analyzed (Participants) | 4 | 5 | 2
  Change from Baselind at D7 | 60.5 (2503.4) | -2179.6 (3108.3) | -1103.3 (168.4)
  Change from Baselind at D10: number analyzed (Participants) | 3 | 5 | 3
  Change from Baselind at D10 | -527.5 (3086.3) | -2066.8 (3342.9) | -1295.0 (359.8)
  Change from Baseline at D13: number analyzed (Participants) | 4 | 5 | 3
  Change from Baseline at D13 | -823.1 (2792.5) | -1931.1 (3601.8) | -1260.6 (781.7)
  Change from baseline at D15 | -506.6 (2518.2) | -2045.2 (3627.7) | -842.6 (1020.0)

5. Secondary Outcome: Change From Baseline in Lactate Dehydrogenase (LDH)
Description: Measured in local units
Time Frame: Baseline, Days 4, 7, 10, 13 and 15
Population: Change from baseline at Days 4, 7, 10, 13 and 15 Data not available for all patients at all timepoints
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
U/L
  Change from Baseline at D4: number analyzed (Participants) | 4 | 5 | 6
  Change from Baseline at D4 | -128.3 (160.9) | -31.8 (13.0) | -70.4 (85.5)
  Change from Baseline at D7: number analyzed (Participants) | 4 | 5 | 4
  Change from Baseline at D7 | -164.3 (267.4) | -16.8 (162.9) | -96.0 (107.3)
  Change from Baseline at D10: number analyzed (Participants) | 4 | 5 | 4
  Change from Baseline at D10 | -184.3 (200.2) | -60.4 (76.4) | -143.5 (128.7)
  Change from Baseline at D13: number analyzed (Participants) | 4 | 5 | 4
  Change from Baseline at D13 | -185.3 (260.9) | -2.6 (264.4) | -155.0 (121.0)
  Change from Baseline at D15 | -163.6 (252.4) | -20.6 (274.8) | -158.4 (108.3)

6. Secondary Outcome: Change From Baseline in D-dimers
Description: Measured in local units
Time Frame: Baseline, Days 4, 7, 10, 13 and 15
Population: Change from baseline at Days 4, 7, 10, 13 and 15 Data not available for all patients at all timepoints
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
nmol/L
  Change from Baseline at D4: number analyzed (Participants) | 5 | 5 | 5
  Change from Baseline at D4 | -0.19 (0.34) | 5.13 (14.73) | -2.05 (1.65)
  Change from Baseline at D7: number analyzed (Participants) | 4 | 5 | 3
  Change from Baseline at D7 | -7.37 (13.84) | 6.78 (19.41) | -4.30 (1.96)
  Change from Baseline at D10: number analyzed (Participants) | 4 | 5 | 3
  Change from Baseline at D10 | -10.07 (18.16) | 4.66 (12.82) | -7.18 (5.96)
  Change from Baseline at D13: number analyzed (Participants) | 4 | 5 | 4
  Change from Baseline at D13 | -7.99 (13.40) | 6.84 (19.39) | -5.67 (7.11)
  Change from Baseline at D15 | -6.84 (12.67) | 6.64 (19.51) | -5.55 (6.45)

7. Secondary Outcome: Change From Baseline in Resting Peripheral Capillary Oxygen Saturation (SpO2)
Description: Measured in percent (%)
Time Frame: Baseline, 3 assessments every Days 4, 7, 10, 13 and 15
Population: Change from baseline at Days 4, 7, 10, 13 and 15 Data not available for all patients at all timepoints
Measure: Mean (Standard Deviation); unit: SpO2%
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
SpO2%
  Change from baseline at D4 | -0.667 (3.598) | 0.267 (2.060) | 0.722 (2.603)
  Change from baseline at D7: number analyzed (Participants) | 4 | 5 | 5
  Change from baseline at D7 | 0.867 (2.923) | 0.667 (1.748) | 2.000 (2.415)
  Change from baseline at D10: number analyzed (Participants) | 4 | 5 | 5
  Change from baseline at D10 | 0.625 (3.523) | 0.267 (1.754) | 2.333 (3.528)
  Change from baseline at D13 | 1.358 (2.140) | -2.233 (6.098) | 1.600 (3.639)
  Change from baseline at D15 | -1.640 (3.383) | -2.400 (5.771) | 2.944 (2.840)

8. Secondary Outcome: Change From Baseline in Oxygen Supplementation
Description: Measured in l/min
Time Frame: Baseline, Days 4, 7, 10, 13 and 15.
Population: Change from baseline at Days 4, 7, 10, 13 and 15 Data not available for all patients at all timepoints
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 4 | 6
L/min
  Change from baseline at D4 | 0.0 (0.0) | 2.8 (5.5) | -0.2 (9.5)
  Change from baseline at D7: number analyzed (Participants) | 4 | 4 | 5
  Change from baseline at D7 | -1.0 (5.8) | -1.8 (4.8) | -7.8 (9.1)
  Change from baseline at D10: number analyzed (Participants) | 4 | 4 | 5
  Change from baseline at D10 | -3.3 (6.9) | -2.3 (6.2) | -17.8 (18.2)
  Change from baseline at D13 | -4.3 (8.1) | -3.3 (7.8) | -20.0 (17.0)
  Change from baseline at D15 | -3.6 (9.3) | -4.3 (7.9) | -15.3 (19.3)

9. Secondary Outcome: Change From Baseline in Partial Pressure of Oxygen/Fraction of Inspired Oxygen (PaO2/FiO2)
Description: Measured in mmHg
Time Frame: Baseline, Day 15
Population: Change from baseline at Day 15 Data not available for the whole population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 2 | 1 | 4
mmHg | 28.98 (106.66) | 51.19 | 156.72 (113.53)

10. Secondary Outcome: Number of Participants With Changes in High-resolution Computed Tomography (CT) Scan of the Chest
Description: Measured in scan evaluation: Normal, Abnormal but not clinically significant, Abnormal clinical significant, Not Done
Time Frame: Screening, Day 15
Population: Data not available for all patients
Measure: Count of Participants; unit: Participants
Groups:
- Emapalumab: Emapalumab i.v. infusion every 3rd day for a total 5 infusions. Day 1: 6mg/kg. Days 4, 7, 10 and 13: 3 mg/kg
  Emapalumab: I.v. infusion every third day
  Abnormal CS at screening
- Anakinra: Anakinra i.v. infusion four times daily for 15 days. 400 mg/day in total, divided into 4 doses given every 6 hours
  Anakinra: Daily i.v. infusion
  Abnormal CS at screening
- Standard of Care: Standard of care according to local practice
  Abnormal CS at screening
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 4 | 4 | 4
Participants
  Normal | 0 | 0 | 1
  Abnormal (NC) | 1 | 3 | 1
  Abnormal (CS) | 3 | 1 | 2

11. Secondary Outcome: Overall Survival
Description: Confirmation of death
Time Frame: Weeks 6 and 10
Measure: Count of Participants; unit: Participants
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
Participants | 2 | 1 | 0

12. Secondary Outcome: Number of Patients With Hospital Discharge
Description: Measured in number of patients
Time Frame: Until discharge up to Week 10
Population: Hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
Participants
  Hospital Discharge | 3 | 4 | 5
  Terminated prior to discharge | 2 | 1 | 1

13. Secondary Outcome: Change of Carbon Dioxide Tension (pCO2) in Hemogasanalysis From Baseline
Description: Measured in local units
Time Frame: Baseline, Days 4, 7, 10, 13 and 15
Population: Change from baseline at Days 4, 7, 10, 13 and 15 Data not available for all patients at all timepoints
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
mmHg
  Change from baseline at D4: number analyzed (Participants) | 3 | 3 | 4
  Change from baseline at D4 | 0.00 (7.21) | -1.00 (3.46) | 2.00 (5.77)
  Change from baseline at D7: number analyzed (Participants) | 3 | 2 | 5
  Change from baseline at D7 | -0.33 (9.45) | 1.00 (1.41) | 5.46 (5.68)
  Change from baseline at D10: number analyzed (Participants) | 3 | 3 | 5
  Change from baseline at D10 | 2.33 (6.03) | 3.67 (8.08) | 4.20 (5.12)
  Change from baseline at D13: number analyzed (Participants) | 2 | 2 | 4
  Change from baseline at D13 | 0.30 (9.48) | 6.50 (3.54) | 0.25 (4.11)
  Change from baseline at D15: number analyzed (Participants) | 3 | 5 | 5
  Change from baseline at D15 | 0.77 (8.33) | 3.75 (5.74) | 4.00 (5.10)

14. Secondary Outcome: Change of Oxygen Tension (pO2) in Hemogasanalysis From Baseline
Description: Measured in local units
Time Frame: Baseline, Days 4, 7, 10, 13 and 15
Population: Change from baseline at Days 4, 7, 10, 13 and 15 Data not available for all patients at all timepoints
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
mmHg
  Change from baseline at D4: number analyzed (Participants) | 3 | 3 | 4
  Change from baseline at D4 | 19.33 (44.28) | 40.67 (34.78) | 5.75 (16.92)
  Change from baseline at D7: number analyzed (Participants) | 3 | 2 | 5
  Change from baseline at D7 | 19.33 (36.56) | 18.50 (13.44) | 23.64 (35.04)
  Change from baseline at D10: number analyzed (Participants) | 3 | 3 | 5
  Change from baseline at D10 | 4.00 (37.36) | -1.33 (11.93) | 4.00 (43.73)
  Change from baseline at D13: number analyzed (Participants) | 2 | 2 | 4
  Change from baseline at D13 | 18.00 (84.85) | -12.00 (5.66) | 24.25 (36.04)
  Change from baseline at D15: number analyzed (Participants) | 3 | 3 | 4
  Change from baseline at D15 | 17.57 (61.05) | 8.75 (47.84) | 8.80 (21.37)

15. Secondary Outcome: Change of Potassium in Hemogasanalysis From Baseline
Description: Measured in local units
Time Frame: Baseline, Days 4, 7, 10, 13 and 15
Population: Change from baseline at Days 4, 7, 10, 13 and 15 Data not available for all patients at all timepoints
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
mmol/L
  Change from baseline at D4: number analyzed (Participants) | 2 | 2 | 2
  Change from baseline at D4 | 0.55 (0.92) | -0.35 (0.49) | 0.45 (1.34)
  Change from baseline at D7: number analyzed (Participants) | 2 | 1 | 4
  Change from baseline at D7 | 0.45 (1.20) | 0.40 | 0.53 (0.93)
  Change from baseline at D10: number analyzed (Participants) | 2 | 2 | 3
  Change from baseline at D10 | 0.25 (0.92) | 0.25 (0.49) | 0.43 (1.22)
  Change from baseline at D13: number analyzed (Participants) | 1 | 1 | 2
  Change from baseline at D13 | -0.50 | 0.10 | 0.10 (0.85)
  Change from baseline at D15: number analyzed (Participants) | 3 | 4 | 4
  Change from baseline at D15 | 0.00 (0.71) | 0.03 (0.75) | 0.17 (0.47)

16. Secondary Outcome: Change of Sodium in Hemogasanalysis From Baseline
Description: Measured in local units
Time Frame: Baseline, Days 4, 7, 10, 13 and 15
Population: Change from baseline at Days 4, 7, 10, 13 and 15 Data not available for all patients at all timepoints
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
mmol/L
  Change from baseline at D4: number analyzed (Participants) | 2 | 2 | 2
  Change from baseline at D4 | 3.0 (5.7) | -0.5 (2.1) | -4.5 (2.1)
  Change from baseline at D7: number analyzed (Participants) | 2 | 1 | 3
  Change from baseline at D7 | 1.0 (1.4) | -5.0 | 0.3 (4.0)
  Change from baseline at D10: number analyzed (Participants) | 2 | 2 | 3
  Change from baseline at D10 | 2.0 (4.2) | -3.0 (7.1) | 1.3 (1.2)
  Change from baseline at D13: number analyzed (Participants) | 1 | 1 | 2
  Change from baseline at D13 | -2.0 | -6.0 | -1.0 (1.4)
  Change from Baseline at D15: number analyzed (Participants) | 2 | 3 | 3
  Change from Baseline at D15 | 2.5 (6.4) | 0.0 (2.6) | 0.7 (2.1)

17. Secondary Outcome: Change of Chloride in Hemogasanalysis From Baseline
Description: Measured in local units
Time Frame: Baseline, Days 4, 7, 10, 13 and 15
Population: Change from baseline at Days 4, 7, 10, 13 and 15 Data not available for all patients at all timepoints
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
mmol/L
  Change from baseline at D4: number analyzed (Participants) | 2 | 2 | 2
  Change from baseline at D4 | 2.0 (5.7) | -0.5 (2.1) | 1.5 (2.1)
  Change from baseline at D7: number analyzed (Participants) | 2 | 1 | 2
  Change from baseline at D7 | 0.5 (0.7) | -4.0 | 2.5 (0.7)
  Change from baseline at D10: number analyzed (Participants) | 2 | 2 | 2
  Change from baseline at D10 | 0.0 (2.8) | -4.5 (3.5) | 4.0 (1.4)
  Change from baseline at D13: number analyzed (Participants) | 1 | 1 | 1
  Change from baseline at D13 | -1.0 | -4.0 | 3.0
  Change from baseline at D15: number analyzed (Participants) | 2 | 3 | 2
  Change from baseline at D15 | 2.0 (4.2) | -2.0 (3.0) | 3.0 (2.8)

18. Secondary Outcome: Change of Lactic Acid in Hemogasanalysis From Baseline
Description: Measured in local units
Time Frame: Baseline, Days 4, 7, 10, 13 and 15
Population: Change from baseline at Days 4, 7, 10, 13 and 15 Data not available for all patients at all timepoints
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
mmol/L
  Change from baseline at D4: number analyzed (Participants) | 1 | 2 | 2
  Change from baseline at D4 | 0.20 | 0.00 (0.28) | -0.45 (1.20)
  Change from baseline at D7: number analyzed (Participants) | 1 | 1 | 2
  Change from baseline at D7 | 0.70 | 1.80 | 0.00 (0.85)
  Change from baseline at D10: number analyzed (Participants) | 1 | 2 | 3
  Change from baseline at D10 | 0.90 | 1.20 (0.17) | -0.50 (0.28)
  Change from baseline at D13: number analyzed (Participants) | 0 | 1 | 1
  Change from baseline at D13 |  | 0.10 | 0.20
  Change from baseline at D15: number analyzed (Participants) | 1 | 3 | 2
  Change from baseline at D15 | 0.00 | 1.27 (1.16) | -0.05 (0.07)

19. Secondary Outcome: Change of Hemoglobin in Hemogasanalysis From Baseline
Description: Measured in local units
Time Frame: Baseline, Days 4, 7, 10, 13 and 15
Population: Change from baseline at Days 4, 7, 10, 13 and 15 Data not available for all patients at all timepoints
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
g/L
  Change from baseline at D4: number analyzed (Participants) | 2 | 2 | 2
  Change from baseline at D4 | -34.0 (46.7) | -15.5 (10.6) | 8.0 (2.8)
  Change from baseline at D7: number analyzed (Participants) | 2 | 1 | 3
  Change from baseline at D7 | -41.0 (65.1) | 3.0 | 6.7 (1.5)
  Change from baseline at D10: number analyzed (Participants) | 2 | 2 | 3
  Change from baseline at D10 | -34.0 (62.2) | 7.5 (6.4) | -1.7 (9.5)
  Change from baseline at D13: number analyzed (Participants) | 1 | 1 | 2
  Change from baseline at D13 | -73.0 | 2.0 | -6.5 (20.5)
  Change from baseline at D15: number analyzed (Participants) | 2 | 3 | 3
  Change from baseline at D15 | -38.0 (49.5) | -3.0 (18.0) | -4.0 (15.9)

20. Secondary Outcome: Change From Baseline in White Blood Cells With Differential Counts
Description: Measured in local units
Time Frame: Baseline, Days 4, 7, 10, 13 and 15
Population: Change from baseline at Days 4, 7, 10, 13 and 15 Data not available for all patients at all timepoints
Measure: Mean (Standard Deviation); unit: 10^9 cells /L
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
10^9 cells /L
  Change from baseline at D4 | 1.000 (4.408) | 0.294 (0.886) | 0.332 (3.009)
  Change from baseline at D7: number analyzed (Participants) | 4 | 5 | 5
  Change from baseline at D7 | 0.340 (2.623) | 2.812 (2.953) | 1.738 (4.165)
  Change from baseline at D10: number analyzed (Participants) | 4 | 5 | 5
  Change from baseline at D10 | 2.728 (1.867) | 4.796 (3.091) | 0.806 (3.643)
  Change from baseline at D13: number analyzed (Participants) | 4 | 5 | 5
  Change from baseline at D13 | 1.548 (5.265) | 1.588 (2.653) | -0.318 (4.079)
  Change from baseline at D15 | 1.686 (4.395) | 1.070 (2.420) | 1.878 (4.788)

21. Secondary Outcome: Change From Baseline in Red Blood Counts
Description: Measured in local units
Time Frame: Baseline, Days 4, 7, 10, 13 and 15
Population: Change from baseline at Days 4, 7, 10, 13 and 15 Data not available for all patients at all timepoints
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
10^12 cells/L
  Change from baseline at D4 | -0.260 (0.470) | -0.022 (0.351) | -0.108 (0.359)
  Change from baseline at D7: number analyzed (Participants) | 4 | 5 | 5
  Change from baseline at D7 | -0.385 (0.732) | 0.016 (0.422) | -0.196 (0.465)
  Change from baseline at D10: number analyzed (Participants) | 4 | 5 | 5
  Change from baseline at D10 | -0.415 (0.875) | 0.220 (0.435) | -0.262 (0.549)
  Change from baseline at D13: number analyzed (Participants) | 4 | 5 | 5
  Change from baseline at D13 | -0.350 (1.254) | 0.106 (0.395) | -0.275 (0.564)
  Change from baseline at D15 | -0.510 (0.969) | 0.004 (0.531) | -0.163 (0.571)

22. Secondary Outcome: Change From Baseline in Hemoglobin
Description: Measured in local units
Time Frame: Baseline, Days 4, 7, 10, 13 and 15
Population: Change from baseline at Days 4, 7, 10, 13 and 15 Data not available for all patients at all timepoints
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
g/L
  Change from baseline at D4 | -6.2 (14.6) | 0.8 (7.0) | -3.5 (9.1)
  Change from baseline at D7: number analyzed (Participants) | 4 | 4 | 5
  Change from baseline at D7 | -9.3 (21.3) | 0.8 (13.1) | -6.2 (10.7)
  Change from baseline at D10: number analyzed (Participants) | 4 | 5 | 5
  Change from baseline at D10 | -11.3 (24.5) | 6.6 (11.9) | -8.0 (16.0)
  Change from baseline at D13: number analyzed (Participants) | 4 | 5 | 5
  Change from baseline at D13 | -10.8 (36.8) | 2.8 (13.6) | -8.2 (17.3)
  Change from baseline at D15 | -14.0 (28.8) | 0.00 (15.6) | -3.7 (16.9)

23. Secondary Outcome: Change From Baseline in Platelet Count
Description: Measured in local units
Time Frame: Baseline, Days 4, 7, 10, 13 and 15
Population: Change from baseline at Day 15 Data not available for all patients at all timepoints
Measure: Mean (Standard Deviation); unit: 10^9 cells /L
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
10^9 cells /L
  Change from baseline at D4 | 29.0 (77.2) | 85.4 (76.7) | 9.8 (153.7)
  Change from baseline at D7: number analyzed (Participants) | 4 | 5 | 5
  Change from baseline at D7 | 19.8 (116.6) | 140.4 (191.8) | 47.4 (232.9)
  Change from baseline at D10: number analyzed (Participants) | 4 | 5 | 5
  Change from baseline at D10 | -3.8 (142.5) | 129.8 (223.9) | 9.0 (232.8)
  Change from baseline at D13: number analyzed (Participants) | 4 | 5 | 5
  Change from baseline at D13 | -32.0 (126.5) | 80.8 (213.2) | -53.8 (191.9)
  Change from baseline at D15 | -37.6 (129.0) | 41.2 (169.3) | -67.2 (158.1)

24. Secondary Outcome: Change From Baseline in Fibrinogen
Description: Measured in local units
Time Frame: Baseline, Days 4, 7, 10, 13 and 15
Population: Change from baseline at Days 4, 7, 10, 13 and 15 Data not available for all patients at all timepoints
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
umol/L
  Change from baseline at D4: number analyzed (Participants) | 5 | 5 | 5
  Change from baseline at D4 | -1.435 (3.137) | -2.434 (1.830) | -0.088 (4.582)
  Change from baseline at D7: number analyzed (Participants) | 4 | 5 | 5
  Change from baseline at D7 | -3.925 (6.113) | -4.898 (2.610) | -1.147 (7.883)
  Change from baseline at D10: number analyzed (Participants) | 4 | 5 | 5
  Change from baseline at D10 | -3.535 (8.998) | -4.980 (2.625) | -5.562 (5.089)
  Change from baseline at D13: number analyzed (Participants) | 4 | 5 | 5
  Change from baseline at D13 | -2.587 (9.308) | -6.227 (2.627) | -5.479 (5.027)
  Change from baseline at D15 | -0.588 (9.210) | -6.380 (2.357) | -4.596 (5.624)

25. Secondary Outcome: Change From Baseline in Complement Factors C3/C4
Description: Measured in local units
Time Frame: Day 15
Population: Change from baseline at Day 15
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
g/L
  C3 | 0.054 (0.094) | -0.068 (0.222) | -0.020 (0.581)
  C4 | 0.024 (0.043) | -0.108 (0.080) | -0.007 (0.192)

26. Secondary Outcome: Change From Baseline in Prothrombin Time
Description: Measured in local units
Time Frame: Baseline, Days 4, 7, 10, 13 and 15
Population: Change from baseline at Day 15 Data not available for all patients at all timepoints
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 4 | 2 | 2
sec
  Change from baseline at D4: number analyzed (Participants) | 3 | 2 | 2
  Change from baseline at D4 | -0.867 (0.058) | 0750 (0.071) | -0.550 (1.344)
  Change from baseline at D7: number analyzed (Participants) | 2 | 2 | 1
  Change from baseline at D7 | -1.250 (0.071) | 0.300 (0.283) | -2.100
  Change from Baseline at D10: number analyzed (Participants) | 3 | 2 | 1
  Change from Baseline at D10 | -1.003 (0.895) | -0.150 (0.919) | -1.700
  Change from Baseline at D13: number analyzed (Participants) | 2 | 2 | 1
  Change from Baseline at D13 | -2.250 (0.354) | 0.050 (0.495) | -1.600
  Change from baseline at D15 | -1.278 (1.087) | -0.150 (0.778) | -0.800 (1.697)

27. Secondary Outcome: Change From Baseline in Cardiac Troponin
Description: Measured in local units
Time Frame: Baseline, Days 4, 7, 10, 13 and 15
Population: Change from baseline at Day 15 Data not available for the whole population
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 1 | 0 | 2
ug/L
  Change from Baseline at D4 | -0.017 |  | 0.002 (0.002)
  Change from Baseline at D7 | -0.022 |  | 0.001 (0.001)
  Change from Baseline at D10 | -0.022 |  | -0.001 (0.001)
  Change from Baseline at D13 | -0.021 |  | -0.001 (0.001)
  Change from Baseline at D15 | -0.022 |  | -0.001 (0.001)

28. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase (AST)
Description: Measured in local units
Time Frame: Baseline, Days 4, 7, 10, 13 and 15
Population: Change from baseline at Day 15 Data not available for all patients at all timepoints
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
U/L
  Change from baseline at D4: number analyzed (Participants) | 4 | 5 | 5
  Change from baseline at D4 | -46.0 (79.8) | -19.2 (32.0) | -63.2 (146.0)
  Change from Baseline at D7: number analyzed (Participants) | 4 | 5 | 5
  Change from Baseline at D7 | -52.8 (107.0) | -27.6 (36.8) | -65.4 (171.1)
  Change from Baseline at D10: number analyzed (Participants) | 4 | 5 | 5
  Change from Baseline at D10 | -53.3 (108.6) | -27.8 (32.9) | -79.8 (170.6)
  Change from Baseline at D13: number analyzed (Participants) | 4 | 5 | 5
  Change from Baseline at D13 | -44.0 (119.3) | -25.2 (28.9) | -83.6 (163.2)
  Change from baseline at D15 | -35.4 (105.3) | -25.8 (28.3) | -77.7 (151.0)

29. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (ALT)
Description: Measured in local units
Time Frame: Baseline, Days 4, 7, 10, 13 and 15
Population: Change from baseline at Day 15 Data not available for all patients at all timepoints
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
U/L
  Change from Baseline D4: number analyzed (Participants) | 4 | 5 | 5
  Change from Baseline D4 | -74.8 (152.9) | 2.6 (38.8) | -23.6 (148.8)
  Change from Baseline D7: number analyzed (Participants) | 4 | 5 | 5
  Change from Baseline D7 | -97.5 (237.1) | 16.6 (66.9) | -62.0 (251.3)
  Change from Baseline D10: number analyzed (Participants) | 4 | 5 | 5
  Change from Baseline D10 | -107.8 (258.3) | 5.0 (54.5) | -107.0 (350.0)
  Change from Baseline D13: number analyzed (Participants) | 4 | 5 | 5
  Change from Baseline D13 | -111.0 (293.3) | -4.8 (51.9) | -119.2 (352.2)
  Change from Baseline at D15 | -90.6 (260.7) | -5.8 (53.2) | -121.8 (309.1)

30. Secondary Outcome: Change From Baseline in Total Bilirubin Levels
Description: Measured in local units
Time Frame: Baseline, Days 4, 7, 10, 13 and 15
Population: Change from baseline at Day 15 Data not available for all patients at all timepoints
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
umol/L
  Change from Baseline at D4: number analyzed (Participants) | 5 | 5 | 5
  Change from Baseline at D4 | -0.171 (3.519) | -1.129 (12.314) | 0.376 (2.600)
  Change from Baseline D7: number analyzed (Participants) | 4 | 5 | 5
  Change from Baseline D7 | -1.496 (4.011) | -0.376 (15.492) | 0.684 (9.922)
  Change from Baseline D10: number analyzed (Participants) | 4 | 5 | 5
  Change from Baseline D10 | -0.385 (4.598) | 4.685 (21.108) | 0.787 (11.931)
  Change from Baseline D13: number analyzed (Participants) | 4 | 5 | 5
  Change from Baseline D13 | -1.710 (4.413) | 13.885 (30.276) | 3.591 (14.146)
  Change from Baseline at D15 | -3.523 (4.473) | 14.125 (29.771) | -0.057 (9.046)

31. Secondary Outcome: Change From Baseline in C-Reactive Protein
Description: Measured in local units
Time Frame: Baseline, Days 4, 7, 10, 13 and 15
Population: Change from baseline at Day 15. Data not available for the whole population
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
mg/L
  Change from Baseline D4: number analyzed (Participants) | 4 | 5 | 4
  Change from Baseline D4 | -53.73 (98.88) | -20.66 (22.29) | -12.65 (12.81)
  Change from Baseline D7: number analyzed (Participants) | 4 | 5 | 4
  Change from Baseline D7 | -63.65 (101.74) | -19.20 (30.95) | -10.98 (19.57)
  Change from Baseline D10: number analyzed (Participants) | 4 | 5 | 4
  Change from Baseline D10 | -60.05 (106.21) | -20.70 (30.57) | -14.60 (15.72)
  Change from Baseline D13: number analyzed (Participants) | 4 | 5 | 4
  Change from Baseline D13 | -60.50 (106.66) | -8.26 (50.51) | -16.33 (14.27)
  Change from Baseline D15: number analyzed (Participants) | 5 | 5 | 5
  Change from Baseline D15 | -38.96 (103.48) | -8.32 (50.53) | -15.26 (12.71)

32. Secondary Outcome: Change From Baseline in Creatinine
Description: Measured in local units
Time Frame: Baseline, Days 4, 7, 10, 13 and 15
Population: Change from baseline at Day 15 Data not available for all patients at all timepoints
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Emapalumab | Anakinra | Standard of Care
Number analyzed (Participants) | 5 | 5 | 6
umol/L
  Change from Baseline D4 | -6.542 (9.430) | 1.414 (8.516) | -6.041 (8.148)
  Change from Baseline D7: number analyzed (Participants) | 4 | 5 | 5
  Change from Baseline D7 | -8.840 (14.454) | 0.530 (6.893) | 0.000 (6.156)
  Change from Baseline D10: number analyzed (Participants) | 4 | 5 | 5
  Change from Baseline D10 | -7.514 (14.481) | 0.000 (5.830) | -0.530 (5.506)
  Change from Baseline D13: number analyzed (Participants) | 4 | 5 | 5
  Change from Baseline D13 | -5.304 (20.171) | 0.000 (8.928) | -1.945 (3.088)
  Change from Baseline D15 | -9.901 (19.281) | -0.354 (9.756) | -5.746 (24.292)

ADVERSE EVENTS:
Time Frame: All fatal and life-threatening SAEs occurring after study drug initiation and up to the end of study visit (Visit 9, Week 10) were reported. All adverse event data were collected from Day 1 to follow-up Week 10.
Arm/Group | Emapalumab | Anakinra | Standard of Care
All-Cause Mortality (participants affected / at risk) | 2/5 | 1/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/5 | 1/5 | 0/6
Other Adverse Events (participants affected / at risk) | 1/5 | 1/5 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emapalumab (N=5) | Anakinra (N=5) | Standard of Care (N=6)
End-stage respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) — Respiratory failure
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) — Respiratory failure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emapalumab (N=5) | Anakinra (N=5) | Standard of Care (N=6)
Atrial Fibrillation (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) — Atrial fibrillation
Muscle Hematoma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Haematoma muscle
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) — Thrombocytopenia
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) — Hypertransaminasaemia two fold increased value

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT04324021/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT04324021/SAP_001.pdf